CLINICAL TRIAL: NCT04183374
Title: DNA Damage and Subfertility in Males - Lifestyle Interventions to Improve Male Fertility and Health
Acronym: ReproDNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regionshospitalet Viborg, Skive (Other)
Responsible Party: Principal Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFI2019Skiveintervention
Record Dates: First submitted 2019-11-08; First posted 2019-12-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Infertility
Keywords: male infertility; DNA fragmentation Index; DFI; life style intervention
MeSH Terms: conditions — Infertility; Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Lifestyle intervention i.e. diet, exercise, smoking cessation, alcohol limitations, dietary supplementation
  Interventions: Other: Life style

INTERVENTIONS:
Other: Life style — Lifestyle intervention i.e. diet, exercise, smoking cessation, alcohol limitations, dietary supplementation

SUMMARY:
A lifestyle intervention study in infertile males of couples seeking fertility treatment with a DNA fragmentation index (DFI) above 15 percentage. A reduction in DNA fragmentation index of 10 percentage points is expected after 3-4 months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* DNA fragmentation index above 15 %

Exclusion Criteria:

* TESA/PESA

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in DNA fragmentation index (DFI) | 3-4 months after inclusion
  DFI is measured by SCSA

SECONDARY OUTCOMES:
Change in classical sperm parameters | 3-4 months after inclusion
  Sperm count
Change in classical sperm parameters | 3-4 months after inclusion
  Sperm motility (movement)
Change in classical sperm parameters | 3-4 months after inclusion
  Sperm morphology (structure)
Change in classical sperm parameters | 3-4 months after inclusion
  Sperm concentration in mio sperm pr. milliliter
Changes in parameters for metabolic syndrome | 3-4 months after inclusion
  Weight in kilograms
Changes in parameters for metabolic syndrome | 3-4 months after inclusion
  Blood pressure in millimeters of mercury
Changes in parameters for metabolic syndrome | 3-4 months after inclusion
  Hemoglobin A1c in mmol/L
Changes in parameters for metabolic syndrome | 3-4 months after inclusion
  Body mass index in kg/m^2
Change in plasma lipids | 3-4 months after inclusion
  Plasma lipids i.e. Total cholesterol, high density lipoprotein, low density lipoprotein and triglycerides
Change in serum D-vitamin levels | 3-4 months after inclusion
  25-hydroxy vitamin D (D3+D2) measured as nmol/l
Number of participants achieving live birth | Week 30-42 of pregnancy
  Birth of a living child after week 23. Registered through self-reported schemes sent to the clinic.
Number of participants with clinical pregnancy | Week 7-8 of pregnancy
  Measurement of heart beat by ultrasound scan
Number of participants with biochemical pregnancy | Day 14-17 of pregnancy
  Increase in serum hCG levels
Cumulative live birth rate | 9-24 months after inclusion
  Live births originating from one controlled stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic Skive, Skive Regional Hospital, Skive, Denmark

IPD SHARING:
Plan to Share IPD: No